CLINICAL TRIAL: NCT04794348
Title: A Phase 2, Multisite, Double-Blind, Prospective Randomized, Crossover, Adequate and Well-Controlled Clinical Trial Assessing the Non-Inferiority of Autologous Freeze Dried Plasma (FDP) to Fresh Frozen Plasma (FFP) in Reversing the Anticoagulation Effects of Warfarin in Healthy Volunteers
Brief Title: Clinical Trial Assessing Non-Inferiority of Freeze Dried Plasma to Fresh Frozen Plasma in Reversing Warfarin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was never started and is no longer planned for execution. We are now in the process of aligning to a new study design with the FDA.
Sponsor: Vascular Solutions LLC (Industry)
Collaborators: United States Army Medical Materiel Development Activity (U.S. Federal Agency); Westat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-18-04
Record Dates: First submitted 2021-03-05; First posted 2021-03-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Anticoagulant Reversal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fresh Frozen Plasma (FFP) (Active Comparator): Subjects will undergo plasmapheresis to generate approximately 1200 mL of fresh frozen plasma. After completion of warfarin dosing, approximately 810 mL of fresh frozen plasma will be intravenously administered to the subject.
  Interventions: Biological: Fresh Frozen Plasma (FFP)
- Freeze Dried Plasma (FDP) (Experimental): Subjects will undergo plasmapheresis to generate approximately 1200 mL, that will be manufactured into freeze dried plasma units. After completion of warfarin dosing, approximately 810 mL of freeze dried plasma will be intravenously administered to the subject.
  Interventions: Biological: Freeze Dried Plasma (FDP)

INTERVENTIONS:
Biological: Fresh Frozen Plasma (FFP) — Autologous units of fresh frozen plasma collected from the subject by plasmapheresis
  Arms: Fresh Frozen Plasma (FFP)
Biological: Freeze Dried Plasma (FDP) — Autologous units of freeze dried plasma manufactured from plasma collected from the subject by plasmapheresis
  Arms: Freeze Dried Plasma (FDP)

SUMMARY:
The purpose of this research study is to see how well an experimental freeze dried plasma product, known as FDP, works to reverse the anticoagulation effects of a prescription medication called warfarin sodium (warfarin) compared to a licensed and routinely used plasma product known as fresh frozen plasma (FFP). The study hypothesis is that FDP is not inferior to FFP when used for this purpose.

Enrolled subjects are required to undergo a minimum of 4 plasmapheresis procedures, generating approximately 2,400 mL. Half will be used as FFP and half will be manufactured into FDP.

Each subject will receive a total of 6 autologous units (approximately 1,620 mL) of plasma product over the course of 2 infusion visits (approximately 810 mL per infusion visit) with a 14 day washout period between infusions.

Warfarin will be administered to each subject prior to each infusion visit. Subjects will be randomized to a treatment arm at their first warfarin administration visit leading up to the first infusion. This establishes the sequence of the plasma products to be infused across the 2 infusion visits. Those randomized to receive 3 units of FDP (approximately 810 mL) at the first infusion visit will receive the equivalent dose of FFP at their second infusion visit and vice versa for those randomized to receive 3 units of FFP at the first infusion visit.

FDP and FFP will be infused intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male or non-pregnant/non-breastfeeding female;
2. Males must weigh ≥ 140 and ≤ 250 pounds; females must weigh ≥ 140 and ≤ 220 pounds;
3. Be ≥ 18 and ≤ 65 years of age;
4. Self-report that he or she feels well and healthy;
5. Score ≥ 35 on the Duke Activity Status Index (see Appendix 3);
6. Be eligible to make plasmapheresis donations based on the AABB Full-Length Donor History Questionnaire with the exception that subjects with a history of travel that puts them at risk for Creutzfeldt-Jakob Disease, malaria, West Nile virus, or Zika virus are eligible for this trial;
7. Males who have sex with men (MSM) and are in monogamous sexual relationships will be allowed to donate and participate in the trial. Other MSM relations will require a 3 month deferral period from the last sexual relation.
8. Have read the educational materials about donating plasma and the information provided on diet, alcohol consumption, warfarin use, and restrictions during the trial;
9. Be able and willing to provide written informed consent;
10. Be available for the duration of the trial (approximately 18 to 28 weeks) and able to come to the treatment clinic for scheduled trial visits;
11. Females should either be surgically sterile (hysterectomy or tubal ligation) or should use a highly effective, medically accepted contraceptive regimen. Highly effective methods of birth control are defined as those that result in a lower failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, condoms with spermicide, or vasectomized partner.
12. All females must have a negative pregnancy test prior to enrollment. Post-menopausal females (women over 50 years of age who, in the absence of pregnancy, have a minimum of 2 months without menses) and females who have had a hysterectomy or oophorectomy will not be tested; and
13. Understand the English language.

Exclusion Criteria:

1. Known liver, kidney, cardiovascular, neurologic, gastrointestinal, blood, endocrine/metabolic, autoimmune or pulmonary disease, or untreated hypertension;
2. Cancer of any kind (except basal cell) under treatment or resolved;
3. Known or past coagulopathy conditions;
4. Any medical conditions or medications on the American Association of Blood Banks (AABB) medical deferral list;
5. Past history of asthma (defined as use of a prescribed daily asthma controller medication or required asthma medication in the past 2 weeks);
6. Past diagnosis of stroke, deep vein thrombosis (DVT), venous or arterial thrombosis, blood clots, or transient ischemic attack;
7. Family history of venous or arterial thrombosis before the age of 50 in first-degree relatives (i.e., biological parents, full siblings, and/or children);
8. D-dimer result > 2.0 FEU/mL;
9. Subjects known to be deficient in protein C or protein S, or found to be deficient as assessed by the investigator based on the screening testing;
10. History of diagnosed pathological arrhythmia;
11. Current smoker (defined as having smoked any form of inhalant within the past 6 months);
12. Subjects who are HIV negative and at high risk for contracting HIV who are currently using pre-exposure prophylaxis (PrEP®) as a prevention method;
13. Known HIV or acquired immunodeficiency syndrome-related illness or received a positive test result for HIV infection;
14. Positive test for hepatitis B virus, hepatitis C virus, human T-cell lymphotropic virus (HTLV), West Nile virus, Zika virus, or syphilis;
15. History of significant treated or untreated mental health issues;
16. Female subject who is pregnant, lactating, or with a positive pregnancy test;
17. Currently taking an antibiotic or another medication for an infection;
18. Treatment or use of aspirin (or other platelet-inhibiting agents) within 14 days of trial donation and infusion visits;
19. Currently using any medications for anticoagulant therapy;
20. Currently using any medications for antiplatelet therapy;
21. Positive urine drug screen for one or more of the following: cannabinoids, cocaine, amphetamines, opiates, or PCP;
22. Previous use of clotting factor concentrate(s);
23. Receipt of blood or blood products within the past 12 months;
24. In the past week, has had a headache and fever at the same time;
25. Known intolerance to any excipients (citrate) in the investigational drug formulation. Intolerance is defined as any subject who exhibits severe symptoms of hypocalcemia after several blood donations;
26. Systolic blood pressure > 140 mm Hg;
27. Diastolic blood pressure > 90 mm Hg;
28. Temperature > 100°F;
29. Known hematocrit ≤ 39% for male donors and ≤ 38% for female donors;
30. Positive direct antiglobulin test (DAT);
31. Treatment with any investigational agent within 1 month before treatment infusion for this trial;
32. Participation in any phase of any other investigational trials while participating in this trial;
33. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule;
34. Other unspecified reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment;
35. Institutionalized because of legal or regulatory order;
36. Follows vegetarian or vegan diet; or
37. Genetically predisposed to be resistant or highly sensitive to warfarin as indicated by having the extensive metabolizer genotypes, VKORC1 missense mutations and/or CYP2C9 variant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Relative change in International Normalized Ratio (INR) | pre-infusion baseline, 6 hours post infusion
  Relative change in INR between pre-infusion baseline and the lowest INR recovery value measured within 6 hours post infusion using equivalent 3-unit doses of FDP compared to FFP
Occurrence of treatment emergent adverse events (TEAE) | Start of first plasma infusion through 14 day follow up visit post second plasma infusion
  Conclusions about safety will be based on the occurrence of TEAEs

SECONDARY OUTCOMES:
Changes in INR | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in aPTT | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in Factor II (FII) | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in Factor VII (FVII) | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in Factor IX (FIX) | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in Factor X (FX) | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in protein C | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Changes in protein S | pre-infusion baseline, 6 hours post infusion
  changes between pre-infusion baseline and 6 hours post-infusion after infusion with FDP compared to FFP
Factor VII (FVII) kinetics area under the curve (AUC) | pre-infusion baseline, 6 hours post infusion
  the AUC for FVII between pre-infusion baseline and 6 hours post infusion with equivalent 3 -unit doses (approximately 810 mL) of FDP vs FFP.
Factor VII (FVII) kinetics maximum concentration (Cmax) | pre-infusion baseline, 6 hours post infusion
  the Cmax for FVII between pre-infusion baseline and 6 hours post infusion with equivalent 3 -unit doses (approximately 810 mL) of FDP vs FFP.
Factor VII (FVII) kinetics half-life (t1/2) | pre-infusion baseline, 24 hours post infusion
  the t1/2 for FVII between pre-infusion baseline and 24 hours post infusion with equivalent 3 unit doses (approximately 810 mL) of FDP vs FFP
Thrombin generation assay (TGA) | 1 hour post infusion
  Report and describe thrombin generation assay (TGA) results after infusion with FDP compared to FFP including lag time, peak amount, and ETP

CONTACTS AND LOCATIONS:
Locations (1):
- Hoxworth Blood Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No